CLINICAL TRIAL: NCT06438315
Title: SuperSaturated Oxygen Comprehensive Observational Registry
Acronym: SSCORE
Status: Recruiting | Type: Observational
Sponsor: TherOx (Industry)
Responsible Party: Sponsor
Other Study IDs: EDC-5731
Record Dates: First submitted 2024-05-21; First posted 2024-05-31 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-12

CONDITIONS: STEMI - ST Elevation Myocardial Infarction; AMI
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- SuperSaturated Oxygen (SSO2) Therapy: Treated with SSO2
  Interventions: Other: No intervention
- Control: Not treated with SSO2
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
The SuperSaturated Oxygen Comprehensive Observational Registry (SSCORE) registry, a prospectively designed observational study, aims to evaluate the clinical utility and effectiveness of SuperSaturated Oxygen (SSO2) Therapy versus percutaneous coronary intervention (PCI) alone among patients with anterior acute myocardial infarction (AMI) in routine clinical practice. The goal is to collect real-world data from patients treated with SSO2 Therapy to determine its impact on the overall heart failure (HF) burden on patients and healthcare systems compared with usual care for treatment of patients with AMI. The SSCORE Registry will generate effectiveness and healthcare resource utilization data that will be used in cost-effectiveness analysis modeling.

ELIGIBILITY:
Inclusion Criteria

Subjects screened for either the Prospective Control Cohort or the SSO2 Treated (On-Label or All Others) Cohorts must meet ALL the following baseline criteria:

* Men or women aged 18 years or older
* Presentation with AMI and successful revascularization of the infarct-related artery with PCI
* The subject or their legally authorized representative has been informed of the nature of the study, agrees to its provisions and has been provided and signed written informed consent, approved by the appropriate Institutional Review Board (IRB)

Treatment with SSO2 Therapy will be up to the physician's discretion and the decision will be made prior to enrollment in the study. Any subject that is treated with SSO2 Therapy and meets the baseline criteria should be invited to participate in the study.

Subjects who are in the Prospective Control Cohort as well as subjects enrolled in the SSO2 Treated On-Label Cohort must meet these additional criteria:

* The primary culprit lesion must be in the left anterior descending (LAD) coronary tree
* Successful primary PCI within 6 hours of symptom onset, as documented by <50% diameter residual angiographic stenosis and Thrombolysis in Myocardial Infarction (TIMI) Grades 2 or 3 flow in the target vessel
* No major complications such as perforation, serious bleeding, or cardiogenic shock
* Not pregnant or nursing

Exclusion Criteria

* Subjects will be excluded if they meet any of the following criteria:
* Life expectancy of less than 2 years
* No access to medical records from either the index hospitalization or subsequent outpatient visits
* Currently participating in an investigational drug or device trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will aim to prospectively enroll 500 subjects not treated with SuperSaturated Oxygen (SSO2) Therapy (Prospective Control Cohort), 500 subjects who received SSO2 Therapy in accordance with the product label (SSO2 Treated On-Label) and any subjects that receive SSO2 at an institution that meet criteria inclusion/exclusion (IE) criteria.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-08-13 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2029-03-31 (Estimated)

PRIMARY OUTCOMES:
Cardiovascular (CV) death or Heart Failure (HF) burden at 1 year | 1 year
  Rate of composite of CV death, new onset HF, any new inpatient or outpatient treatment for HF, or worsening of HF

SECONDARY OUTCOMES:
Time to Cardiovascular (CV) death or HF burden | 2 years
  Days to the composite of CV death, new onset HF, any new inpatient or outpatient treatment for HF, or worsening of HF
Rate of all cause mortality | 2 years
  Rate of all cause mortality
Rate of All-cause Hospitalization | 2 years
  Rate of All-cause Hospitalization
Rate of cardiovascular death | 2 years
  Rate of cardiovascular death
Rate of Hospitalization for Heart Failure | 2 years
  Rate of Hospitalization for Heart Failure
Major Adverse Cardiovascular Events (MACE) | 2 years
  composite of rates of CV death, reinfarction, or HF hospitalization
Rate of Reinfarction | 2 years
  Rate of Reinfarction
Change in EQ5D-3L Score | 2 years
  Patient reported outcome, 0 to1, where 0 is death and 1 is perfect health
Change in Kansas City Cardiomyopathy Questionnaire (KCCQ-23) Score | 2 years
  Heart related patient reported outcome, scaled from 0 to 100, with 0 representing the worst symptoms and function and 100 representing the best
Change in % of Left ventricular ejection fraction (LVEF) | 2 years
  Rate of change of LVEF from baseline to time point
Change in New York Heart Association (NYHA) classification scale, I-IV | 2 years
  Rate of change of NHYA classification from baseline to time point

CONTACTS AND LOCATIONS:
Overall Officials: William W O'Neill, MD, Principal Investigator — Henry Ford Hospital
Locations (22):
- United States (22):
  - MemorialCare Orange Coast Medical Center, Fountain Valley, California
  - UCSD Health La Jolla - Sulpizio Cardiovascular Center, La Jolla, California
  - MemorialCare Saddleback Medical Center, Laguna Hills, California
  - MemorialCare Long Beach Medical Center, Long Beach, California
  - UCSD Hillcrest Medical Center, San Diego, California
  - Baptist Health Baptist Hospital, Miami, Florida
  - NCH Baker Hospital, Naples, Florida
  - NCH North Naples, Naples, Florida
  - University of Chicago, Chicago, Illinois
  - Carle Health Methodist Hospital, Peoria, Illinois
  - Ascension Via Christi St Francis, Wichita, Kansas
  - Corewell Health Dearborn Hospital, Dearborn, Michigan
  - Mercy Hospital, Coon Rapids, Minnesota
  - Abbott Northwestern Hospital, Minneapolis, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - North Shore University Hospital, Manhasset, New York
  - Long Island Jewish Hospital, Queens, New York
  - Charleston Area Medical Center, Charleston, West Virginia
  - St Mary's Medical Center, Huntington, West Virginia
  - Aurora St Luke's Medical Center, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stone GW, Martin JL, de Boer MJ, Margheri M, Bramucci E, Blankenship JC, Metzger DC, Gibbons RJ, Lindsay BS, Weiner BH, Lansky AJ, Krucoff MW, Fahy M, Boscardin WJ; AMIHOT-II Trial Investigators. Effect of supersaturated oxygen delivery on infarct size after percutaneous coronary intervention in acute myocardial infarction. Circ Cardiovasc Interv. 2009 Oct;2(5):366-75. doi: 10.1161/CIRCINTERVENTIONS.108.840066. Epub 2009 Sep 15. PMID 20031745
- [Background] David SW, Khan ZA, Patel NC, Metzger DC, Wood FO, Wasserman HS, Lotfi AS, Hanson ID, Dixon SR, LaLonde TA, Genereux P, Ozan MO, Maehara A, Stone GW. Evaluation of intracoronary hyperoxemic oxygen therapy in acute anterior myocardial infarction: The IC-HOT study. Catheter Cardiovasc Interv. 2019 Apr 1;93(5):882-890. doi: 10.1002/ccd.27905. Epub 2018 Sep 28. PMID 30265429